CLINICAL TRIAL: NCT00862238
Title: An Arts Intervention for Drug-Using Homeless Youth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Adeline Nyamathi, MD, Distinguished Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 081101501; 1R21DA023521 (NIH)
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Drug Use
MeSH Terms: interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Art Messaging (Experimental): 4-session educational group which utilizes art, photography, film, painting to portray a message to reduce drug use, and prevent hepatitis A, B, & C
  Interventions: Behavioral: Art Messaging
- Health Promotion (Other): 4-session education offering basic information about the prevention of hepatitis A, B & C
  Interventions: Other: Health Promotion

INTERVENTIONS:
Behavioral: Art Messaging — 4-session educational group which utilizes art, photography, film, painting to portray a message to reduce drug use, and prevent hepatitis A, B, & C
  Arms: Art Messaging
Other: Health Promotion — 4 session education which offers basic information about the prevention of hepatitis A, B, & C
  Arms: Health Promotion

SUMMARY:
In the study, homeless youth from a drop-in site and faculty from UCLA and California Institute of the Arts will develop, pilot test and evaluate a youth-based drug and health-promoting program. It is hoped that this program will help in the development of a program that can be further tested in a larger study and lead to the development of an innovative and effective drug counseling program that youth situated in homeless sites will utilize.

DETAILED DESCRIPTION:
Nationwide, homeless youths are attempting to escape major life challenges, which may result in problem drug and alcohol use. Such behaviors are associated with hepatitis virus infections and HIV. Less than one third of homeless youth seek medical care, and less than 10% of drug and alcohol-using youths seek substance abuse treatment services. Based upon increasing knowledge about the barriers experienced by homeless youth relating to accessing treatment for substance use and health promoting services, it is clear that homeless youth need to play a major role in the planning, implementation and evaluation of drug counseling programs delivered at sites that homeless youth frequent. Using a community-based participatory research (CBPR) approach, UCLA researchers recently engaged homeless youth and community partners in qualitative research to better understand homeless youths' perspectives on drug counseling and to consider innovative strategies to engage homeless youth, in accessing drug use and health promotion counseling. Our community partners included homeless youth from homeless youth-based organizations, and faculty from the California Institute of the Arts (CalArts). An innovative youth-centered strategy considered by homeless youth was the use of the arts and media to craft personal messages that capture youth interest and appeal. In the proposed investigation, researchers, homeless youth and staff from a drop-in site frequented by homeless youth, along with our CalArts partners, will participate in the development, pilot testing and evaluation of a youth-centered drug-use and health-promoting intervention program. In Phase I of this R21, a CBPR approach will be utilized with a steering committee to develop a youth-centered drug use and health promoting intervention program, LIFE MATTERS which will be assessed in terms of acceptability via focus group sessions with street youth and subsequently refined based upon homeless youth feedback. In Phase 2, investigators and community partners will conduct a pilot study to explore the acceptability of the LIFE MATTERS program as well as test the impact of the program, compared to a control group, with 80 similar youth in terms of: completion of the program; reduction of risky drug and alcohol use; completion of a HAV/HBV vaccine series; and improvement in knowledge about hepatitis. The short-term goals are to refine strategies that can be fully tested in a large-scale intervention trial. The long-term goals are to contribute to knowledge about promoting innovative and youth-designed drug-related behaviors, and treatment completion in settings where youth congregate.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for this Phase II study of 128 homeless youth recruited from Common Ground (described in Phase I) include:

  1. unsheltered homeless, 15-24 years of age, and frequenting the study site;
  2. screened as a moderate-to-heavy drug user;
  3. willing to be tested for HAV/HBV at baseline; and
  4. not a participant of the Phase I study.

Exclusion Criteria:

* Cognitively impaired and not a participant of Phase I.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2008-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Conduct a pilot study to explore the acceptability of the LIFE-MATTERS program, and estimate the impact of the program, compared to the control group. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Common Ground, Santa Monica, California, United States